CLINICAL TRIAL: NCT04180410
Title: Monitoring of Regional Lung Ventilation by Chest Electrical Impedance in the Course of Extubation
Acronym: EXIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A02986-51
Record Dates: First submitted 2019-11-24; First posted 2019-11-27 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: No-randomized,no-comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EIT (Other): Electrical Impedance Tomography is performed before extubation, during follow up visits of extubation and 48H after extubation
  Interventions: Device: EIT

INTERVENTIONS:
Device: EIT — Electrical Impedance Tomography is performed before extubation, during follow-up visits of extubation and 48H after extubation. Follow-up visits are shortened in case of extubation failure.

SUMMARY:
The Electrical Impedance Tomography (EIT) is a non-invasive exam. This exam performed on the lung continuously produces cross-sectional images of lung function. It may be relevant in lung description.

DETAILED DESCRIPTION:
The aim is to follow the patients after extubation for the lung description.

EIT exam is performed before extubation, during follow-up visits and 48H after extubation

ELIGIBILITY:
Inclusion Criteria:

1. Age> 65 years
2. Invasive mechanical ventilation time greater than 48 hours
3. known or suspected Chronic obstructive pulmonary disease
4. Known or suspected heart failure
5. Success in the spontaneous ventilation and extubation test scheduled by the doctor in charge
6. Patient or trusted person who has been informed of the study and has consented to participate

Exclusion Criteria:

1. Pregnant women, minor patients
2. Patients under extracorporeal circulatory assistance (ECMO)
3. Refusal of the patient
4. Contraindications to the realization of the phrenic nerve stimulation technique:

   * Pacemaker, implantable cardiac defibrillator and other pacemakers
   * Spinal implants, thoracic drains ...
   * Copper allergy
   * Epileptic patients
5. Patients performing uncontrolled body movements
6. Contraindications to the realization of the technique of Electrical Imaging Tomography:

   * Breast circumference not between 70 cm and 150 cm.
   * Body mass index (BMI) greater than 50
   * Impossibility of placing the CT belt at the level of the chest skin (lesions, bandages, dressings, chest drains ...)
   * Patients with unstable spinal lesions or fractures
   * Allergy to tomography belt materials: silicone, brass, stainless steel
   * Pacemaker, implantable cardiac defibrillator and other pacemakers
7. Patients under legal protection (tutorship / guardianship)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-08-19 (Estimated); Study Completion 2021-08-19 (Estimated)

PRIMARY OUTCOMES:
acute respiratory failure | 48 hours
  Occurrence of extubation failure

SECONDARY OUTCOMES:
pulmonary ventilation | 48 hours
  lung pulmonary volume (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Aphp_La Pitie Salpetriere, Paris, France

REFERENCES:
- [Derived] Joussellin V, Bonny V, Spadaro S, Clerc S, Parfait M, Ferioli M, Sieye A, Jalil Y, Janiak V, Pinna A, Dres M. Lung aeration estimated by chest electrical impedance tomography and lung ultrasound during extubation. Ann Intensive Care. 2023 Sep 26;13(1):91. doi: 10.1186/s13613-023-01180-3. PMID 37752365